CLINICAL TRIAL: NCT01570504
Title: Randomized, Open-label, Multi Centre Phase III Clinical Trial on Multiple Versus Single Dose of Ivermectin for the Treatment of Strongyloidiasis
Brief Title: Multiple Versus Single Dose of Ivermectin for the Treatment of Strongyloidiasis
Acronym: STRONGTREAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro per le Malattie Tropicali (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTD1-2012; 2011-002784-24 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-04-04 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Strongyloidiasis
Keywords: Strongyloidiasis; Strongyloides stercoralis; Ivermectin
MeSH Terms: conditions — Strongyloidiasis | interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ivermectin multiple doses (Experimental): A dose of 200 mcg/kg of ivermectin given on days 1,2, 15 and 16
  Interventions: Drug: Ivermectin
- 1 dose ivermectin (Active Comparator): A single 200 mcg/kg dose of ivermectin
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Ivermectin — oral formulation
  Other Names: Stromectol

SUMMARY:
Ivermectin is currently the best drug to cure strongyloidiasis, but the "standard" single dose of 200 mcg/kg is probably not enough to guarantee cure. As strongyloidiasis can be fatal in immunosuppressed patients, it is mandatory to define the optimal dosage to eradicate the parasite.

Aim of this study is to define the most effective dose schedule of ivermectin to cure strongyloidiasis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients older than 5 years and weighting > 15 kg
* Current residence in non-endemic areas
* Either direct diagnosis of S. stercoralis infection AND positive serology at any titer OR positive serology at "high" titer, irrespective of results of direct tests

Exclusion Criteria:

* Pregnant or lactating women
* Subjects suffering from CNS diseases
* Disseminated strongyloidiasis
* Immunocompromised patients.
* Lack of informed consent
* Previous treatment with ivermectin (in the last year)

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
clearance of strongyloides infection | 12 months
  Clearance of infection is defined by: negative stool agar/charcoal culture/RT-PCR - direct examination of three faecal samples for S. stercoralis AND negative serology or decrease in titer below a defined cutoff

SECONDARY OUTCOMES:
All-cause mortality during the 12 months of follow-up. | 12 months
Patients with partial response to treatment at T 2 | 12 months
Patients with adverse reactions | From Day 1st to Day 5th of treatment and from Day 15th to Day 19th (or 72 hours from treatment completion)
  grade 1 to 5 as defined in detailed protocol
Patients with increase in blood ALT over cutoff value | Day 17
Patients with decrease in WBC count below cutoff value | Day 17
Average difference in blood ALT and WBC count at day 17, compared with baseline | Day 17
Average difference in blood eosinophil count at T2, compared with baseline | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zeno Bisoffi, MD, PhD, Principal Investigator — Centre for Tropical Diseases, Negrar (Verona), Italy
Locations (9):
- Italy (4):
  - Centro per le Malattie Tropicali, Ospedale Sacro Cuore, Negrar, Verona
  - Clinica di Malattie Infettive e Tropicali, Brescia
  - UFDID, Azienda Ospedaliero-universitaria Careggi, Florence
  - Unità di Malattie Infettive, Anna Meyer Children's Universisty Hospital, Florence
- Spain (3):
  - Unidad de Medicina, Hospital de Poniente-El Ejido, El Ejido, Almeria
  - FCRB, Hospital Clinic de Barcelona, Barcelona
  - Unitat Medicina Tropical i Salut Internacional Drassanes, Barcelona
- United Kingdom (2):
  - Addenbrookes Hospital, Cambridge University Hospital, Cambridge
  - UCLH, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buonfrate D, Salas-Coronas J, Munoz J, Maruri BT, Rodari P, Castelli F, Zammarchi L, Bianchi L, Gobbi F, Cabezas-Fernandez T, Requena-Mendez A, Godbole G, Silva R, Romero M, Chiodini PL, Bisoffi Z. Multiple-dose versus single-dose ivermectin for Strongyloides stercoralis infection (Strong Treat 1 to 4): a multicentre, open-label, phase 3, randomised controlled superiority trial. Lancet Infect Dis. 2019 Nov;19(11):1181-1190. doi: 10.1016/S1473-3099(19)30289-0. Epub 2019 Sep 23. PMID 31558376